CLINICAL TRIAL: NCT05739630
Title: An Multicenter, Randomized, Controlled, Prospective Clinical Study of Mitoxantrone Liposome Combined With PTCy as Conditioning Regimen in Allo-HSCT in Acute Leukemia
Brief Title: M-PTCy vs BuCy in Haploidentical HSCT for Acute Leukemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023003
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M+PTCy group (Experimental): For the M-PTCy group, Mitoxantrone liposomes with 36mg/m2 and Bu 3.2mg/kg -5 to -4, Flu 30mg/m2 -12 to -9, Ara-C 1.5g/m2 -12 to -9，CTX 15mg/kg/d -3 to -2, was used as conditioning regimen, Post Transplant Cyclophosphamide 50 mg/kg IV daily on days +3 and +4.
  Interventions: Drug: mitoxantrone liposome
- BuCy group (Active Comparator): For the BUCY group, the conditioning regimen involved Ara-C 2g/m2 q12h -8, BU 3.2 mg/kg -7 to -5,CTX 1.8 g/m2 -4 to -3, to prevent GVHD, MTX 15mg/m2 +1d, 10mg/m2 +3,+6,+11,CsA 3mg/kg/d from -8d,MMF 1g q12h from -8d， ATG 2.5mg/kg/d -5 to -2.
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: mitoxantrone liposome — Mitoxantrone liposomes with 36mg/m2 and Bu 3.2mg/kg -5 to -4, Flu 30mg/m2 -12 to -9, Ara-C 1.5g/m2 -12 to -9，CTX 15mg/kg/d -3 to -2, was used as conditioning regimen, Post Transplant Cyclophosphamide 50 mg/kg IV daily on days +3 and +4.
  Other Names: Fludarabine,Cytarabine,busulfan,Cyclophosphamide,MMF,Tacrolimus Capsules
  Arms: M+PTCy group
Drug: ATG — Control group:the conditioning regimen involved Ara-C 2g/m2 q12h -8, BU 3.2 mg/kg -7 to -5,CTX 1.8 g/m2 -4 to -3, to prevent GVHD, MTX 15mg/m2 +1d, 10mg/m2 +3,+6,+11,CsA 3mg/kg/d from -8d,MMF 1g q12h from -8d， ATG 2.5mg/kg/d -5 to -2.
  Other Names: MECCNU,Hu,Cytarabine,busulfan,Cyclophosphamide,MTX,CsA
  Arms: BuCy group

SUMMARY:
This study intends to evaluate the efficiency and safety of M-PTCy as conditioning regimen in Haploidentical HSCT for Acute Leukemia, so as to provide a new conditioning regimen for allogeneic hematopoietic cell transplantation.

DETAILED DESCRIPTION:
Haploidentical related donor transplantation is now considered an important alternative to allogeneic hematopoietic stem cell transplantation (allo-HSCT). Posttransplant cyclophosphamide (PTCy) has revolutionized Haplo HCT with acceptable rates of engraftment, graft-versus-host disease (GVHD), relapse, and survival.To prolonger PFS, OS and alleviate GVHD, we combined Mitoxantrone liposomes with PTCy as conditioning regimen in allogeneic hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. The patients meet the diagnostic criteria for acute leukemia(except APL).
2. Expecting life span is more than 3 months.
3. The patients intended allogeneic hematopoietic stem cell transplantation.

Exclusion Criteria:

1. Previously received doxorubicin or other anthracycline therapy, the total cumulative dose of doxorubicin≥360 mg/m2.
2. Cardiac function and disease meet one of the following conditions:

   1. Long QTc syndrome or QTc intervalgt≥480 ms;
   2. Complete left bundle branch block, grade II or III Degree atrioventricular block;
   3. Severe, uncontrolled arrhythmia requiring drug treatment;
   4. New York Society of Cardiology class ≥ II;
   5. Cardiac ejection fraction (LVEF) lower than 50% or lower than the study The lower limit of the central laboratory test value range;
   6. History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, clinically serious pericardial disease history within 6 months before recruitment, or ECG evidence of acute ischemia or active conduction system abnormalities.
3. Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN); Total bilirubin > 1.5 times upper limit of normal; Serum creatinine > 1.5 times the upper limit of normal.
4. Suffering from other malignant tumors in the past or at the same time ;
5. Exclude patients with severe active infection or other underlying diseases who cannot tolerate chemotherapy;
6. Human immunodeficiency virus (HIV) infected patients (HIV antibody positive);
7. Active hepatitis B and C infection；
8. Pregnant women, lactating women, and patients who refuse to take effective contraceptive measures during the study;
9. Severe mental disorders who do not cooperate with treatment;
10. Judgment by the investigator , There are patients who are not suitable to participate in this study.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the 1st day to 2 years after enrollment
  It is defined as the total survival of a patient after CR until the tumor recurrence or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | From the 1st day to 2 years after enrollment
  The time from randomization to death from any cause.
incidence of GVHD | From the 1st day to 2 years after enrollment
  The incidence of graft-versus-host disease
CMV and EBV activation | From the 1st day to 2 years after enrollment
  The incidencance of cytomegalovirus and Epstein-barr virus infection

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, MD/phD, Principal Investigator — Study Principle investigator
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Apperley J, Niederwieser D, Huang XJ, Nagler A, Fuchs E, Szer J, Kodera Y. Reprint of: Haploidentical Hematopoietic Stem Cell Transplantation: A Global Overview Comparing Asia, the European Union, and the United States. Biol Blood Marrow Transplant. 2016 Mar;22(3 Suppl):S15-8. doi: 10.1016/j.bbmt.2016.01.006. PMID 26899273